CLINICAL TRIAL: NCT02410018
Title: An Open Label, Single Center, Pilot Study to Evaluate the Safety and Effectiveness of OCL 503 in the Treatment of Women With Leiomyomata Scheduled for Hysterectomy
Brief Title: Safety and Effectiveness of OCL 503 in the Treatment of Women With Leiomyomata
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IMBiotechnologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCL503-P1-UFE-01
Record Dates: First submitted 2015-03-06; First posted 2015-04-07 (Estimated); Results first posted 2018-09-07 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Leiomyomata
MeSH Terms: interventions — Uterine Artery Embolization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 - Uterine Artery Embolization (Experimental): Women treated with OCL 503 proceeding to hysterectomy 1 week post embolization.
  OCL 503 will be administered by catheter to the uterine artery(ies) to achieve blood flow stasis.
  Interventions: Device: OCL 503 (uterine artery embolization)
- Cohort 2 - Uterine Artery Embolization (Experimental): Women treated with OCL 503 proceeding to hysterectomy 1 month post embolization.
  OCL 503 will be administered by catheter to the uterine artery(ies) to achieve blood flow stasis.
  Interventions: Device: OCL 503 (uterine artery embolization)

INTERVENTIONS:
Device: OCL 503 (uterine artery embolization) — Transcatheter embolization of the uterine artery(ies) using an embolic agent.

SUMMARY:
This is a prospective, pilot, open-label, uncontrolled, safety and effectiveness study of uterine artery embolization with OCL 503 in women with leiomyomata who are scheduled for hysterectomy.

DETAILED DESCRIPTION:
Patients will be allocated to Cohort 1 or Cohort 2. Following pelvic angiogram to delineate the uterine vasculature, embolization procedures of the left and right uterine arteries (as required) will be performed on each patient, using OCL 503 as the embolic agent. Patients in Cohort 1 will proceed to hysterectomy 1 week after embolization, and patients in Cohort 2 will undergo hysterectomy 1 month after embolization. Tumor response, as measured by changes in leiomyomata size and perfusion, will be determined by Magnetic Resonance Imaging or Magnetic Resonance Angiography. Histology of the resected uterus will be conducted to evaluate inflammatory response and viable tumour tissue.

ELIGIBILITY:
Inclusion Criteria:

* presence of one or more of the following symptoms: abnormal menstrual bleeding, prolonged menstrual period, pelvic pain, or bulk-related symptoms that are attributed to uterine fibroids (bulk-related symptoms include pelvic pressure, abdominal distension, abdominal bloating, constipation, backache, urinary frequency, urinary retention, ureteral dilation, and rectal pressure), and the intensity of uterine fibroid-related symptoms, which are sufficiently sever to warrant hysterectomy, and the patient's medical history, physical examination, and the results of imaging by ultrasound or MRI;
* are between the ages of 30 and 55 years, inclusive;
* have had a pelvic examination by a gynaecologist within the previous 6 months;
* have had a normal Pap smear within the last 12 months;
* have had an endometrial biopsy within the previous three to six months, as appropriate to patient history;
* are premenopausal with menstrual cycles lasting between 22 and 35 days. A follicle stimulating hormone (FSH) value obtained within three months prior to the procedure must be < 40 IU/L;
* are scheduled for total abdominal hysterectomy;
* are willing and able to provide written, informed consent.

Exclusion Criteria:

* have been treated with gonadotropin-releasing hormone (GnRH) agonists within the previous 12 weeks;
* have a American Society of Anesthesiologists (ASA) score ≥ 3;
* have abnormally large ovarian arteries, as assessed by MRA and determined by the Investigator;
* have an undiagnosed pelvic mass outside the uterus;
* have claustrophobia or other contraindications to the performance of the pre- and post-procedure MRI studies including the presence of metal implants, metal plates, bone pins, bone screws, neurostimulators, cardiac pacemakers, aneurysm clips, cochlear or retinal implants, permanent hearing aids, or permanent eye-liner;
* have pedunculated subserosal fibroids with an attachment to the uterus less than one third of the greatest diameter of the fibroid;
* who do not agree to use contraceptives from Visit 1 until undergoing total abdominal hysterectomy;
* have compromised hematopoietic function;
* have hepatic dysfunction defined as liver function tests 30% above the upper limit of normal;
* have an active gynecologic or systemic infection;
* have renal dysfunction as defined by a serum creatinine > 1.5 mg/dL
* have a history of gynecologic malignancy;
* have had a documented anaphylactic reaction to a drug or anesthetic, or an allergic reaction to iodine contrast media not controlled by antihistamines or steroids;
* have received other investigational drugs or who have had experimental therapy within the past four weeks or are participating in any other concurrent experimental therapy;
* have a uterine volume < 250 mL or approximately > 24 weeks gestation;
* have known endometrial hyperplasia, adenomyosis, or pelvic inflammatory disease;
* have abnormal coagulation profiles;
* are allergic to bovine collagen;

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Siskin, MD, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical Center, Albany, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 - Uterine Artery Embolization: Women treated with OCL 503 proceeding to hysterectomy 1 week post embolization.
  OCL 503 will be administered by catheter to the uterine artery(ies) to achieve blood flow stasis.
  OCL 503 (uterine artery embolization): Transcatheter embolization of the uterine artery(ies) using an embolic agent.
- Cohort 2 - Uterine Artery Embolization: Women treated with OCL 503 proceeding to hysterectomy 1 month post embolization.
  OCL 503 will be administered by catheter to the uterine artery(ies) to achieve blood flow stasis.
  OCL 503 (uterine artery embolization): Transcatheter embolization of the uterine artery(ies) using an embolic agent.
Period: Overall Study
Arm/Group | Cohort 1 - Uterine Artery Embolization | Cohort 2 - Uterine Artery Embolization
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Uterine Artery Embolization | Cohort 2 - Uterine Artery Embolization | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events
Description: Short-term safety of OCL 503 at 7 days post treatment of women with leiomyomata by UAE, as measured by Adverse Events reporting - Serious Adverse Events
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Uterine Artery Embolization | Cohort 2 - Uterine Artery Embolization
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

2. Primary Outcome: Change in Fibroid Perfusion From Baseline at 7 Days Post Treatment
Description: Number of participants with decreased fibroid perfusion from baseline at 7 days post treatment of women with leiomyomata by UAE - Decreased Fibroid Perfusion Fibroid perfusion indicative of blood flowing to the fibroid at baseline and 7 days after embolization was determined using MRI.
Time Frame: Baseline and 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Uterine Artery Embolization | Cohort 2 - Uterine Artery Embolization
Number analyzed (Participants) | 2 | 1
Participants | 2 | 1

3. Primary Outcome: Number of Participants With Serious Adverse Events
Description: Short-term safety of OCL 503 at 28 days post treatment of women with leiomyomata by UAE, as measured by Adverse Events reporting - Serious Adverse Events
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Uterine Artery Embolization | Cohort 2 - Uterine Artery Embolization
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

4. Primary Outcome: Change in Fibroid Perfusion From Baseline at 28 Days Post Treatment of Women With Leiomyomata by UAE
Description: Number of participants with decreased fibroid perfusion from baseline at 28 days post treatment of women with leiomyomata by UAE.
Time Frame: Baseline and 28 days
Population: Decrease in fibroid perfusion
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Uterine Artery Embolization | Cohort 2 - Uterine Artery Embolization
Number analyzed (Participants) | 0 | 1
Participants | 0 | 1

5. Secondary Outcome: Tissue Necrosis Assessed by Histology Graded Scale at 7 Days Post Treatment of Women With Leiomyomata by UAE
Description: Tissue necrosis assessed by histology at 7 days post treatment of women with leiomyomata by UAE - Fibroid necrosis observed
Time Frame: 7 days
Population: Histological assessment of uterine tissue was conducted for Cohort 1 at 7-days, post-embolization. Histological assessment of uterine tissue was conducted for Cohort 2 at 28-days, post-embolization.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Uterine Artery Embolization | Cohort 2 - Uterine Artery Embolization
Number analyzed (Participants) | 2 | 1
Participants | 2 | 0

6. Secondary Outcome: Inflammatory Response Assessed by Histology at 7 Days Post Treatment of Women With Leiomyomata by UAE
Description: Inflammatory response assessed by histology at 7 days post treatment of women with leiomyomata by UAE - Perivascular inflammation - Low Grade
Time Frame: 7 days
Population: Inflammatory response for Cohort 1 was assessed at 7-days, post-embolization. Inflammatory response for Cohort-2 was assessed at 28-days, post-embolization.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Uterine Artery Embolization | Cohort 2 - Uterine Artery Embolization
Number analyzed (Participants) | 2 | 1
Participants | 2 | 0

7. Secondary Outcome: Tissue Necrosis Assessed by Histology Graded Scale at 28 Days Post Treatment of Women With Leiomyomata by UAE
Description: Tissue necrosis assessed by histology graded scale at 28 days post treatment of women with leiomyomata by UAE - Fibroid Necrosis
Time Frame: 28 days
Population: Histological assessment of uterine tissue was conducted at 7-days for Cohort 1 and 28-days for Cohort 2, post-embolization.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Uterine Artery Embolization | Cohort 2 - Uterine Artery Embolization
Number analyzed (Participants) | 2 | 1
Participants | 0 | 1

8. Secondary Outcome: Inflammatory Response Assessed by Histology at 28 Days Post Treatment of Women With Leiomyomata by UAE
Description: Inflammatory response assessed by histology at 28 days post treatment of women with leiomyomata by UAE - Perivascular Low Grade
Time Frame: 28 days
Population: Inflammatory response was conducted at 7-days post-embolization for Cohort 1 and 28-days for Cohort 2, post-embolization.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Uterine Artery Embolization | Cohort 2 - Uterine Artery Embolization
Number analyzed (Participants) | 2 | 1
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Day 0 through 28 days.
Arm/Group | Cohort 1 - Uterine Artery Embolization | Cohort 2 - Uterine Artery Embolization
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Uterine Artery Embolization (N=2) | Cohort 2 - Uterine Artery Embolization (N=1)
Fibroid expulsion (Reproductive system and breast disorders) | 0 (0) | 0 (0) — Expulsion of embolized fibroid from the uterine cavity. Note: risk of this adverse event is lost upon the study subject undergoing standard of care hysterectomy. All study subjects underwent hysterectomy.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Uterine Artery Embolization (N=2) | Cohort 2 - Uterine Artery Embolization (N=1)
Post-embolization Syndrome (Investigations) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No